CLINICAL TRIAL: NCT00970983
Title: Randomized Clinical Trial Comparing Axillary Dissection "by Principle" and Axillary Dissection Based on the Histological Result of the Sentinel Node, in Patients With Breast Carcinoma of Small Size
Brief Title: Axillary Dissection Based on the Histological Result of the Sentinel Node, in Patients With Breast Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO 185
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- QUART (Active Comparator): Patients in this arm will receive quadrantectomy, axillary dissection and radiotherapy (the current standard therapy).
  Interventions: Procedure: quadrantectomy and axillary dissection
- QURT (SN-) (Experimental): Patients will receive quadrantectomy, sentinel node investigation and radiotherapy. Selective axillary dissection will be performed if sentinel node is positive.
  Interventions: Procedure: quadrantectomy + sentinel node biopsy

INTERVENTIONS:
Procedure: quadrantectomy and axillary dissection — standard quadrantectomy and axillary dissection
  Arms: QUART
Procedure: quadrantectomy + sentinel node biopsy — standard quadrantectomy and selective axillary dissection only if sentinel node biopsy is positive
  Arms: QURT (SN-)

SUMMARY:
The purpose of this study is to evaluate the disease free and overall survival of patients with breast carcinomas of small size, i.e., not greater than 2.0 cm and with clinically non palpable axillary lymph nodes, undergoing either conservative surgery and axillary dissection, or a similar treatment for the primary tumor and rapid analysis of the sentinel lymph node, the result of which determines axillary node dissection or its avoidance is based.

DETAILED DESCRIPTION:
The axillary lymph nodes represent the most frequent site of metastasis from breast carcinoma. In previous studies, it has been shown that the process of metastasis to the axillary nodes proceeds in an orderly and progressive fashion from the I to the II and to the III level and that a "saltatory" event of metastasis represents a rare event described in only 2% to 6% of cases.

The risk of metastasis is directly correlated with the size of the primary tumor. When smaller than 1 cm in diameter, the risk of metastasis is about 10%; when larger than 5 cm in diameter, the risk increases to more than 70%.

The involvement of axillary lymph nodes by metastases constitutes today the most important prognostic factor in breast cancer. Massive invasion is most certainly associated with a poor outcome and therefore, the information that the lymph node status can provide, is indispensible for administration of appropriate therapies in the postoperative period. Nevertheless, in those cases where the lymph nodes are found to be free of metastases, axillary dissection is a useless treatment that can prove harmful if one considers all the possible short and long term complications.

Presently, there are no diagnostic modalities that are able to provide an accurate lymph node staging preoperatively. This information can only be gained by histologic examination of all lymph nodes after complete axillary dissection.

Standard treatment for operable breast cancer today always involves the dissection of the axillary lymph nodes, regardless of the surgical procedure used for resection of the primary tumor, i.e. conservative or demolitive. This not only results in a large expenditure of resources (longer surgical procedures under general anesthesia), but most notably, in an increased risk of complications (lymphedema and functional limitations of the involved extremity) for the patient, secondary to a more aggressive intervention on the axilla.

A method utilizing preoperative lymphoscintigraphy and intraoperative use of a gamma-ray probe in order to evaluate the possibility of metastasis in the first axillary lymph node, i.e. the "sentinel node", has recently been put into practice at our institute. This method, which in its first part consists in the subcutaneous or peritumoral administration of a radiolabeled (99Tc) human albumin colloid (see methods section), has allowed isolation and excision of the sentinel lymph node with the use of the gamma-ray probe in 98.8% of cases.

In the case that this procedure should prove highly predictable of patient outcome, numerous axillary lymphadenectomies could be avoided and with such, numerous complications associated with such aggressive intervention.

A first phase study has evaluated 238 patients with breast carcinoma that would be candidates for complete axillary dissection. Patients with intraductal carcinoma, those candidates for primary chemotherapy, those diagnosed during pregnancy or lactation, and those with tumors less than 1 cm in size (because of inclusion in the randomized trial (053) evaluating the role of radiotherapy on the axilla in patients undergoing conservative surgery without axillary node dissection) were excluded from the study. The results of this first phase have shown a concordance in the histologic findings between the sentinel lymph node and all remaining axillary lymph nodes, subdivided into three levels, in 96.7% of cases. Furthermore, concordance was 100% in 18 patients with breast carcinoma of a size equal or less than 1.0 cm.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years.
* Clinical, mammographic or ultrasonographic diagnosis of a unicentric carcinoma with an ultrasonographic diameter of equal or less than 2.0 cm.
* Although not a factor of exclusion, a breast scintigraphy using MDP-99m is recommended for accurate determination of possible multifocality or multicentricity of the tumor, as well as for the determination of possible bone metastasis.
* Axillary lymph nodes that cannot be palpated or that are not clinically suspicious for metastasis.
* No previously executed therapy (including biopsy) at any outside institution.
* Those patients with nonpalpable lesions will be subjected to preoperative radioactive occult lesion localization (ROLL) or stereotactic biopsy.
* Adequate patient information and signature of the informed consent.

Exclusion Criteria:

* Lesions diagnosed as non-infiltrating (in-situ) ductal or lobular carcinoma.
* Paget's disease.
* Documented multicentricity and/or abundant multifocality of the neoplasm.
* Clinically metastatic lymph nodes.
* Patients previously biopsied at other institutions.
* Carcinomas detected during pregnancy or lactation.
* Histotypes diverse from breast carcinoma lesions.
* History of previous malignancy (excluding basocellular carcinoma, in-situ cervical carcinoma and/or contralateral breast carcinoma without recurrence for at least 15 years of follow-up).

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 1998-03; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
disease free survival, overall survival | every 6 months for the first 5 years and every 8 months afterwards

SECONDARY OUTCOMES:
number of axillary metastases | every 6 months for the first 5 years and every 8 months afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Veronesi, MD, Study Director — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Milano, Italy

REFERENCES:
- [Derived] Veronesi U, Viale G, Paganelli G, Zurrida S, Luini A, Galimberti V, Veronesi P, Intra M, Maisonneuve P, Zucca F, Gatti G, Mazzarol G, De Cicco C, Vezzoli D. Sentinel lymph node biopsy in breast cancer: ten-year results of a randomized controlled study. Ann Surg. 2010 Apr;251(4):595-600. doi: 10.1097/SLA.0b013e3181c0e92a. PMID 20195151